CLINICAL TRIAL: NCT03370965
Title: Optic Neuritis Differential Diagnosis Study (ONDDS)
Brief Title: Optic Neuritis Differential Diagnosis Study
Acronym: ONDDS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Center of Martinique (Other)
Collaborators: University Hospital Center of Guadeloupe (Unknown); Hospital Center of Cayenne (French Guyana) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17/B/01
Record Dates: First submitted 2017-10-20; First posted 2017-12-13 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Optic Neuritis; Neuromyelitis Optica; Multiple Sclerosis
Keywords: optic neuritis; neuromyelitis optica; multiple sclerosis; emergent treatment of optic neuritis; optic neuritis disease modifying therapy; optic neuritis treatment trial; plasma exchange
MeSH Terms: conditions — Optic Neuritis; Neuromyelitis Optica; Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with optic neuritis (Experimental)
  Interventions: Diagnostic Test: Neuro-ophtalmology examination

INTERVENTIONS:
Diagnostic Test: Neuro-ophtalmology examination — Patients will first undergo a full neuro-ophthalmic examination which includes visual acuity, contrast vision, color vision, slit-lamp anterior segment and fundus examination as well as automatized visual field and optical coherence tomography of the optic nerves and retina.
  Patients will then be admitted to the Neurology and Ophthalmologic Department for optic neuritis emergency treatment, 3-Tesla brain and medullar MRIs, and ancillary testing. Specific NMO antibodies (AQP-4 and MOG) will be tested in all patients. Neuro-ophthalmic examination will be repeated after 3 days of IV steroids in order to decide on further treatment.

SUMMARY:
Background: Optic neuritis is a frequent cause of vision loss encountered by ophthalmologists in the Caribbean. The diagnosis is made on clinical grounds. Optic neuritis can occur either in an isolated manner or, most often, as the first symptom of multiple sclerosis (MS) or neuromyelitisoptica (NMO). These 2 demyelinating disorders differ by many means, including treatment and prognosis. MS can cause severe long-term disability while NMO is a short-term sight- and life-threatening condition causing potential relapses, which may require plasma exchanges. Furthermore, disease-modifying therapies used in NMO are different from those used in MS, which can worsen the natural history of NMO. Early differential diagnosis of these diseases is thus crucial for preventing severe visual loss and disability.

DETAILED DESCRIPTION:
Background: Optic neuritis is a frequent cause of vision loss encountered by ophthalmologists in the Caribbean. The diagnosis is made on clinical grounds. Optic neuritis can occur either in an isolated manner or, most often, as the first symptom of multiple sclerosis (MS) or neuromyelitisoptica (NMO). These 2 demyelinating disorders differ by many means, including treatment and prognosis. MS can cause severe long-term disability while NMO is a short-term sight- and life-threatening condition causing potential relapses, which may require plasma exchanges. Furthermore, disease-modifying therapies used in NMO are different from those used in MS, which can worsen the natural history of NMO. Early differential diagnosis of these diseases is thus crucial for preventing severe visual loss and disability.

Purpose: The investigators aim to identify early predictive factors (clinical, biological and radiological) of NMO occurrence in patients presenting with optic neuritis and with no prior history of demyelinating diseases.

Method: The investigators will conduct a multicentric prospective study including all patients of 18 years or older, with no prior history of demyelinating disorders and presenting with a diagnosis of optic neuritis in Martinique, Guadeloupe, French Guiana, Saint-Martin and Saint-Barthélemy. Patients will first undergo a full neuro-ophthalmic examination which includes visual acuity, contrast vision, color vision, slit-lamp anterior segment and fundus examination as well as automatized visual field and optical coherence tomography of the optic nerves and retina. Patients will then be admitted to the Neurology and Ophthalmologic Department of the University Hospital of Martinique for optic neuritis emergency treatment, 3-Tesla brain and medullar MRIs, and ancillary testing. Specific NMO antibodies (AQP-4 and MOG) will be tested in all patients. Neuro-ophthalmic examination will be repeated after 3 days of IV steroids in order to decide on further treatment. Patients will be further monitored at 1, 6 and 12 months so as to determine the most likely etiology of optic neuritis with the aid of MS and NMO diagnosis criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged 18 years or older at time of inclusion.
2. Table of unilateral or bilateral optic neuritis defined as follows (clinical diagnosis):

   1. Visual sharpness (acuity and / or visual field) experienced acutely or subacutely (<1 month) unilateral or bilateral, not corrected by optical correction.
   2. Absence of ophthalmologic lesion which may explain the visual loss.
   3. Examination of the normal fundus or showing a pallor or papular edema.
   4. Presence of relative pupillary deficit relative if unilateral attack.
3. Patient (s) affiliated to a social security scheme (beneficiary or beneficiary).
4. Patient who has given free and written consent.

Exclusion Criteria:

1. Patients known to have an inflammatory disease of the central nervous system (MS, NMO, EMAD).
2. Known history of inflammatory pathology (lupus or sarcoidosis) or infectious pathology (syphilis, HIV) that may give rise to optical neuropathy.
3. Table suggestive of Leber's hereditary optic neuropathy (genetically confirmed).
4. Treatment in progress known to give optical neuropathies.
5. Consumption of toxic known to give optical neuropathies.
6. Drinking more than 3 alcohol drinks per day for men and 2 alcohol drinks per day for women over a period of more than 15 years.
7. Arguments for non-arteritic ischemic optic neuropathy defined by all of the following criteria:

   1. Absence of pain in eye movements.
   2. Altitudinal deficit of the visual field.
   3. Choroidal ischemia with fluorescein angiography.
   4. Presence of cardiovascular risk factors.
   5. Absence of neurological signs related to inflammatory disease of the central nervous system.
8. Arguments for arterial ischemic optic neuropathy defined by all of the following criteria:

   1. Absence of pain in eye movements.
   2. Altitudinal deficit of the visual field.
   3. Choroidal ischemia with fluorescein angiography.
   4. Presence of symptoms suggestive of Horton's disease.
   5. Absence of neurological signs related to inflammatory disease of the central nervous system.
9. Pregnant and lactating patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-06-07 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Final diagnosis using MS (McDonald, 2010) - Spatial dissemination | 12 months
  One T2 lesion ore more in at least two of the four central nervous system territories considered to be characteristic of MS:
  * juxtacortical,
  * periventricular,
  * sub-tentorial,
  * medullary (in case of medullary syndrome or brain stem, symptomatic lesions are excluded from the diagnostic criteria and do not participate in the lesion count).
Final diagnosis using MS (McDonald, 2010) - Time dissemination | 12 months
  * A new lesion in T2 and / or a lesion taking gadolinium on a follow-up MRI regardless of the time of initial MRI.
  * The simultaneous presence of asymptomatic lesions raised and not elevated by gadolinium at any time.
NMO diagnosis criteria (Wingerchuk, 2015) - Diagnosis of NMO-SD with positive anti-AQP4 Antibody | 12 months
  * At least one main clinical criterion (1)
  * Exclusion of other diagnoses
NMO diagnosis criteria (Wingerchuk, 2015) - Diagnosis of NMO-SD with anti-AQP4 negative antibody | 12 months
  * At least 2 main clinical criteria occurring in the context of one or more clinical outbreaks and meeting the following criteria
    * At least 1 of the 2 main clinical criteria should be optic neuritis, extensive longitudinal myelitis or area postrema syndrome.
    * Dissemination in space (at least 2 main criteria)
    * Respect of MRI imaging criteria (2)
  * Anti-AQP4 negative antibodies
  * Exclusion of differential diagnoses

CONTACTS AND LOCATIONS:
Overall Officials: Philippe CABRE, PhD, Principal Investigator — Centre Hospitalier Universitaire de Martinique
Locations (1):
- CHU of Martinique, Fort-de-France, France

IPD SHARING:
Plan to Share IPD: No